CLINICAL TRIAL: NCT01998607
Title: Survey of Oncology Practitioners Prescribing XGEVA® in Europe to Evaluate Their Knowledge of XGEVA® Summary of Product Characteristics Pertaining to Osteonecrosis of the Jaw
Brief Title: Survey of XGEVA® Presrcibers in Europe to Evaluate Their Knowledge of the Summary of Product Characteristics Pertaining to Osteonecrosis of the Jaw
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20110102
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumours; Bone Metastasis
Keywords: Solid tumours; Bone Metastasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Round 1: Survey of 210 oncologists 12 - 18 months after commercial availability of XGEVA® in the respective country
  Interventions: Other: Physician Survey
- Round 2: Survey of 210 oncologists 24 - 30 months after commercial availability of XGEVA® in the respective country
  Interventions: Other: Physician Survey

INTERVENTIONS:
Other: Physician Survey — Eligible physicians will be contacted to perform the physician survey. A standardised online questionnaire will be used to collect information about the physician's awareness of the Summary of Product characteristics (SPC) pertaining to osteonecrosis of the jaw (ONJ) in the last 6-18 months.
  Other Names: This is an observational study.

SUMMARY:
Osteonecrosis of the Jaw (ONJ) is an adverse effect of antiresorptive therapy that is well-recognized in patients with advanced cancer. Detailed information regarding this risk is specified in the Summary of Product Characteristics (SPC). The statements in the SPC are the most important mechanism for minimizing the risk for ONJ. The study objective is to measure the knowledge of oncology practitioners prescribing XGEVA® regarding the content pertaining to ONJ in the SPC after commercial availability.

DETAILED DESCRIPTION:
This is a multiple cross-sectional survey study of practicing oncology practitioners prescribing XGEVA in Europe from across but not limited to the 5 largest European countries by population (including France, Germany, Italy, Spain and the U.K.) and 4 Nordic countries (Denmark, Finland, Norway and Sweden). The survey will be conducted in two rounds. The two survey rounds will be conducted 12 to 18 months and 24 to 30 months after XGEVA becomes commercially available in the participating countries. The initial contact and screening of potential participating oncology practitioners will continue until a total of 210 eligible and consenting oncology practitioners complete the survey per round. For the 5 largest European countries by population, it is intended that 30 oncology practitioners will be surveyed per country per survey round. If this sample size cannot be achieved, oncology practitioners from another country in that region will be surveyed to achieve a regional sample size of 150 per survey round. Oncology practitioners from the Nordic countries will be surveyed to achieve a regional sample size of 60 per survey round. For all countires, the number of surveys collected in each country in the second survey round will, where possible, equate to the number of surveys collected in each country in the first survey round.

ELIGIBILITY:
Practicing oncology specialists who have treated at least 5 adult patients with bone metastases from solid tumours in the last quarter. Must have prescribed XGEVA® within the last 12 months. Must not have participated in a previous survey round

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Oncology specialists treating adult patients with bone metastases from solid tumours
Sampling Method: Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2013-02-04 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-05-15 (Actual)

PRIMARY OUTCOMES:
Proportion of participating oncology practitioners prescribing XGEVA® who are aware of the SPC statements pertaining to ONJ (each question pertaining to a SPC statement will be assessed seperately at the end of each survey round) | 12 and 24 months after commercial availability of XGEVA® in the respective country

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com